CLINICAL TRIAL: NCT03142451
Title: A Randomized, Multicenter, Double-blind, Vehicle-controlled Study to Evaluate the Safety and Efficacy of FMX103 1.5% Topical Minocycline Foam Compared to Vehicle in the Treatment of Facial Papulopustular Rosacea (FX2016-11)
Brief Title: A Study (Study 1) to Evaluate the Safety and Efficacy of FMX103 1.5% Topical Minocycline Foam in the Treatment of Facial Papulopustular Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FX2016-11
Record Dates: First submitted 2017-04-27; First posted 2017-05-05 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Facial Papulopustular Rosacea
Keywords: Topical Minocycline Foam; 2-Arm study; Inflammatory lesion counts; Investigator's Global Assessment score

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study, with limited access to the randomization code. The randomization code will be held in confidence until after the study database is locked and a memo documenting the database lock has been issued. Every effort will be made to retain the integrity of the blind. When issued to the sites, the study drug will be identical in appearance for all participants, regardless of treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- FMX103 1.5% (Experimental): Participants will apply the assigned FMX103 minocycline foam 1.5% topically once daily for 12 weeks as directed.
  Interventions: Drug: FMX103 minocycline foam 1.5%
- Vehicle foam (Placebo Comparator): Participants will apply the assigned vehicle foam topically once daily for 12 weeks as directed.
  Interventions: Drug: Vehicle foam

INTERVENTIONS:
Drug: FMX103 minocycline foam 1.5% — Dosage form description: Foam containing minocycline HCl 1.5%. Once daily application of a sufficient amount of foam to cover the entire face. Estimated maximum is 0.5 g of drug product containing 7.5 mg (1.5% active) of minocycline. Participants will apply a small amount of the drug as a thin layer over all areas of the face. Participants should apply the drug at approximately the same time each day, about 1 hour before bedtime.
  Arms: FMX103 1.5%
Drug: Vehicle foam — Dosage form description: Foam containing minocycline vehicle foam. Once daily application of a sufficient amount of foam to cover the entire face. Estimated maximum is 0.5 g of drug product containing 0.0 mg (vehicle) of minocycline. Participants will apply a small amount of the drug as a thin layer over all areas of the face. Participants should apply the drug at approximately the same time each day, about 1 hour before bedtime.
  Arms: Vehicle foam

SUMMARY:
The primary objectives of this study are to determine the efficacy and safety of FMX103 1.5% minocycline foam applied topically once daily for 12 weeks in the treatment of rosacea.

DETAILED DESCRIPTION:
This is a randomized, multicenter, double-blind, vehicle-controlled, 2 arm study to evaluate the safety and efficacy of FMX103 topical foam containing 1.5% minocycline compared to vehicle, in the treatment of participants with moderate-to-severe facial papulopustular rosacea. Qualified participants will be randomized in a 2:1 ratio (active:vehicle) to receive 1 of the following 2 treatments:

* FMX103 minocycline foam 1.5%
* Vehicle foam

Participants will be assigned to 1 of 2 treatments according to the randomization schedule. Participants will apply (or have applied) the study drug topically once daily for 12 weeks as directed. Participants will be advised to use the study drug at approximately the same time each day. Both the Investigator and participant will be blinded to the study drug identity. Participants will return for visits at Weeks 1, 4, 6, 8, 10, and 12. Efficacy evaluations (inflammatory lesion counts and Investigator's Global Assessment [IGA] score) will be performed at Weeks 4, 8, and 12 during the study.

Note: Originally the two studies FX2016-11 and FX2016-12 were combinedly presented in the protocol registration form under one NCT number (NCT03142451), and later separated since results were analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate-to-severe rosacea (as per the IGA score) on the proposed facial treatment area consisting of:

   1. At least 15 and not more than 75 facial papules and pustules, excluding lesions involving the eyes and scalp;
   2. No more than 2 nodules on the face.
2. Presence of or history of erythema and/or flushing on the face.

Exclusion Criteria:

1. Presence of any skin condition and/or Excessive facial hair, on the face that would interfere with the diagnosis or assessment of rosacea.
2. Moderate or severe rhinophyma, dense telangiectasia (score 3, severe), or plaque-like facial edema.
3. History of hypersensitivity or allergy to minocycline, any other tetracycline, or of any other component of the formulation.
4. Active ocular rosacea (eg, conjunctivitis, blepharitis, or keratitis) of sufficient severity to require topical or systemic antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (54):
  - Foamix Investigational Site #152, Tucson, Arizona
  - Foamix Investigational Site # 127, Fremont, California
  - Foamix Investigational Site #155, Los Angeles, California
  - Foamix Investigational Site #143, Northridge, California
  - Foamix Investigational Site # 131, Oceanside, California
  - Foamix Investigational Site #156, Oceanside, California
  - Foamix Investigational Site #153, San Diego, California
  - Foamix Investigational Site # 114, San Diego, California
  - Foamix Investigational Site # 116, San Luis Obispo, California
  - Foamix Investigational Site # 135, Santa Ana, California
  - Foamix Investigational Site # 123, Santa Monica, California
  - Foamix Investigational Site # 109, Clearwater, Florida
  - Foamix Investigational Site # 112, Hialeah, Florida
  - Foamix Investigational Site #150, Lake Worth, Florida
  - Foamix Investigational Site #149, Miami, Florida
  - Foamix Investigational Site #151, Miami, Florida
  - Foamix Investigational Site #144, Miami Lakes, Florida
  - Foamix Investigational Site # 104, Ormond Beach, Florida
  - Foamix Investigational Site # 121, Sanford, Florida
  - Foamix Investigational Site #154, Sweetwater, Florida
  - Foamix Investigational Site # 125, Tampa, Florida
  - Foamix Investigational Site # 142, West Palm Beach, Florida
  - Foamix Investigational Site # 124, West Palm Beach, Florida
  - Foamix Investigational Site # 118, Alpharetta, Georgia
  - Foamix Investigational Site # 139, Snellville, Georgia
  - Foamix Investigational Site # 138, New Albany, Indiana
  - Foamix Investigational Site # 102, Metairie, Louisiana
  - Foamix Investigational Site # 115, New Orleans, Louisiana
  - Foamix Investigational Site # 110, Beverly, Massachusetts
  - Foamix Investigational Site # 107, Brighton, Massachusetts
  - Foamix Investigational Site # 137, Ann Arbor, Michigan
  - Foamix Investigational Site # 103, Fort Gratiot, Michigan
  - Foamix Investigational Site # 120, Troy, Michigan
  - Foamix Investigational Site # 140, Warren, Michigan
  - Foamix Investigational Site # 130, Saint Joseph, Missouri
  - Foamix Investigational Site # 133, Omaha, Nebraska
  - Foamix Investigational Site #146, Las Vegas, Nevada
  - Foamix Investigational Site # 136, New York, New York
  - Foamix Investigational Site #145, New York, New York
  - Foamix Investigational Site # 111, Stony Brook, New York
  - Foamix Investigational Site # 119, Charlotte, North Carolina
  - Foamix Investigational Site # 101, Bexley, Ohio
  - Foamix Investigational Site # 128, Dublin, Ohio
  - Foamix Investigational Site #147, Broomall, Pennsylvania
  - Foamix Investigational Site # 141, Jenkintown, Pennsylvania
  - Foamix Investigational Site #157, Saint Clair, Pennsylvania
  - Foamix Investigational Site # 129, Yardley, Pennsylvania
  - Foamix Investigational Site # 105, Johnston, Rhode Island
  - Foamix Investigational Site # 106, Greenville, South Carolina
  - Foamix Investigational Site # 122, Murfreesboro, Tennessee
  - Foamix Investigational Site # 117, Austin, Texas
  - Foamix Investigational Site #159, Houston, Texas
  - Foamix Investigational Site # 108, San Antonio, Texas
  - Foamix Investigational Site # 126, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — http://foamix.co.il/

RESULTS

PARTICIPANT FLOW:
Groups:
- FMX103 1.5%: Participants applied the assigned FMX103 minocycline foam 1.5% topically once daily for 12 weeks as directed.
- Vehicle Foam: Participants applied the assigned vehicle foam topically once daily for 12 weeks as directed.
Period: Overall Study
Arm/Group | FMX103 1.5% | Vehicle Foam
Started | 495 | 256
Completed | 437 | 232
Not Completed | 58 | 24
Not completed — Adverse Event | 5 | 2
Not completed — Lost to Follow-up | 25 | 8
Not completed — Participant request | 24 | 12
Not completed — Protocol Violation | 3 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FMX103 1.5% | Vehicle Foam | Total
Number analyzed (Participants) | 495 | 256 | 751
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (13.71) | 49.7 (12.85) | 49.2 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 355 | 186 | 541
  Male | 140 | 70 | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 165 | 88 | 253
  Not Hispanic or Latino | 328 | 168 | 496
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
  Black or African American | 7 | 4 | 11
  White | 474 | 241 | 715
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Absolute Change From Day 0/Baseline in the Inflammatory Lesion Count at Week 12
Description: To determine the efficacy of FMX103 1.5% minocycline foam applied topically once daily for 12 weeks in the treatment of rosacea. Lesion counts included the number of papules, pustules, and nodules.
  Change from Baseline was calculated as the value at Baseline minus the post-Baseline value. Thus, a positive change reflects a reduction in lesion count.
Time Frame: Baseline and Week 12
Population: The intent-to-treat (ITT) population included all randomized participants. Analyses using the ITT population were based on the randomized treatment.
Measure: Mean (Standard Error); unit: Lesions
Arm/Group | FMX103 1.5% | Vehicle Foam
Number analyzed (Participants) | 495 | 256
Lesions | 17.56 (0.442) | 15.34 (0.604)
Statistical Analysis 1: Comparison: FMX103 1.5% vs Vehicle Foam; Test type: Superiority; p = 0.0031, ANCOVA; Analysis of covariance (ANCOVA) model includes treatment, baseline inflammatory lesion count, and analysis center; Mean Difference (Final Values) = 2.21, 95% CI 2-sided [0.75 to 3.68], Standard Error of Mean 0.749

2. Primary Outcome: Percentage of Participants Achieving Investigator Global Assessments (IGA) Treatment Success at Week 12
Description: To determine the efficacy of FMX103 1.5% minocycline foam applied topically once daily for 12 weeks in the treatment of rosacea. The Investigator assessed the global severity of rosacea using the IGA scale. The scale ranges from 0 (Clear): No inflammatory papules or pustules to 4 (Severe): Many inflammatory papules or pustules, and up to 2 nodules. Higher scores indicated severe outcome. Treatment success was defined as an IGA score of 0 (clear) or 1 (almost clear), and at least a 2-step improvement (decrease) from Day 0/Baseline.
Time Frame: Week 12
Population: The ITT population included all randomized participants. Analyses using the ITT population were based on the randomized treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | FMX103 1.5% | Vehicle Foam
Number analyzed (Participants) | 495 | 256
Percentage of participants | 52.1 | 43.0
Statistical Analysis 1: Comparison: FMX103 1.5% vs Vehicle Foam; Test type: Superiority; p = 0.0273, Cochran-Mantel-Haenszel — The p-value is for the null hypothesis that the combined risk ratio equals 1; Cochran-Mantel-Haenszel Test Stratified by Analysis Center; Risk Ratio (RR) = 1.210, 95% CI 2-sided [1.022 to 1.434]

3. Secondary Outcome: Percentage of Participants Achieving IGA Treatment Success of at Least 2 Grades at Week 12
Description: To determine the efficacy of FMX103 1.5% minocycline foam applied topically once daily for 12 weeks in the treatment of rosacea. The Investigator assessed the global severity of rosacea using the IGA scale. The scale ranges from 0 (Clear): No inflammatory papules or pustules to 4 (Severe): Many inflammatory papules or pustules, and up to 2 nodules. Higher scores indicated severe outcome. Treatment success was defined as a 2-grade improvement (decrease) in score at Week 12 compared to Day 0/Baseline.
  Here, overall number of participants analyzed signifies only the participants with available data that were analyzed for the outcome measure.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | FMX103 1.5% | Vehicle Foam
Number analyzed (Participants) | 423 | 225
Percentage of participants | 55.3 | 45.8
Statistical Analysis 1: Comparison: FMX103 1.5% vs Vehicle Foam; Test type: Superiority; p = 0.0171, Cochran-Mantel-Haenszel — The p-value is for the null hypothesis that the combined risk ratio equals 1; Cochran-Mantel-Haenszel Test Stratified by Analysis Center; Risk Ratio (RR) = 1.210, 95% CI 2-sided [1.028 to 1.425]

4. Secondary Outcome: The Percent Change From Day 0/Baseline in Inflammatory Lesion Count at Week 12
Description: To determine the efficacy of FMX103 1.5% minocycline foam applied topically once daily for 12 weeks in the treatment of rosacea. Lesion counts included the number of papules, pustules, and nodules.
  Here, overall number of participants analyzed signifies only the participants with available data that were analyzed for the outcome measure.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | FMX103 1.5% | Vehicle Foam
Number analyzed (Participants) | 423 | 225
Percent change | 64.13 (1.584) | 56.52 (2.133)
Statistical Analysis 1: Comparison: FMX103 1.5% vs Vehicle Foam; Test type: Superiority; p = 0.0039, ANCOVA; ANCOVA model includes treatment, Baseline inflammatory lesion count, and analysis center; Mean Difference (Final Values) = 7.62, 95% CI 2-sided [2.46 to 12.77], Standard Error of Mean 2.626

5. Secondary Outcome: The Absolute Change From Day 0/Baseline in the Inflammatory Lesion Counts at Week 4 and Week 8
Description: To determine the efficacy of FMX103 1.5% minocycline foam applied topically once daily for 12 weeks in the treatment of rosacea. Lesion counts included the number of papules, pustules, and nodules. The change from Baseline was calculated as the value at Baseline minus the post-Baseline value. Thus, a positive change reflects a reduction in lesion count.
Time Frame: Baseline, Week 4 and Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | FMX103 1.5% | Vehicle Foam
Number analyzed (Participants) | 495 | 256
Lesions
  Week 4 | 11.24 (0.441) | 8.62 (0.608)
  Week 8 | 15.59 (0.445) | 12.51 (0.610)
Statistical Analysis 1: Comparison: FMX103 1.5% vs Vehicle Foam; Statistical analysis for Week 4; Test type: Superiority; p = 0.0004, ANCOVA; ANCOVA model included treatment, Baseline inflammatory lesion count, and analysis center; Mean Difference (Final Values) = 2.63, 95% CI 2-sided [1.16 to 4.09], Standard Error of Mean 0.747
Statistical Analysis 2: Comparison: FMX103 1.5% vs Vehicle Foam; Statistical analysis for Week 8; Test type: Superiority; p < 0.0001, ANCOVA; ANCOVA model included treatment, Baseline inflammatory lesion count, and analysis center; Mean Difference (Final Values) = 3.09, 95% CI 2-sided [1.62 to 4.56], Standard Error of Mean 0.750

6. Secondary Outcome: Percentage of Participants Achieving IGA Treatment Success at Week 4 and Week 8
Description: To determine the efficacy of FMX103 1.5% minocycline foam applied topically once daily for 12 weeks in the treatment of rosacea. The Investigator assessed the global severity of rosacea using the IGA scale. The scale ranges from 0 (Clear): No inflammatory papules or pustules to 4 (Severe): Many inflammatory papules or pustules, and up to 2 nodules. Higher scores indicated severe outcome. Treatment success was defined as an IGA score of 0 (clear) or 1 (almost clear), and at least a 2-grade improvement (decrease) from Day 0/Baseline.
Time Frame: Week 4 and Week 8
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | FMX103 1.5% | Vehicle Foam
Number analyzed (Participants) | 495 | 256
Percentage of participants
  Week 4 | 15.3 | 9.1
  Week 8 | 35.2 | 29.4
Statistical Analysis 1: Comparison: FMX103 1.5% vs Vehicle Foam; Statistical analysis for Week 4; Test type: Superiority; p = 0.0201, Cochran-Mantel-Haenszel — P-value is for the null hypothesis that the risk ratio equals 1; Cochran-Mantel-Haenszel test stratified by analysis center; Risk Ratio (RR) = 1.685, 95% CI 2-sided [1.085 to 2.616]
Statistical Analysis 2: Comparison: FMX103 1.5% vs Vehicle Foam; Statistical analysis for Week 8; Test type: Superiority; p = 0.1278, Cochran-Mantel-Haenszel — P-value is for the null hypothesis that the risk ratio equals 1; Cochran-Mantel-Haenszel test stratified by analysis center; Risk Ratio (RR) = 1.191, 95% CI 2-sided [0.951 to 1.492]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: To evaluate the tolerability and safety of topical minocycline foam applied once daily for 12 weeks. A treatment-emergent adverse events (TEAE) was defined as any AE with an onset date on or after the first application of study drug, and before to the last application of study drug plus 3 days, having been absent pre-treatment or worsening relative to the pre-treatment state.
Time Frame: From Day 0/Baseline until the Safety Follow-up (4 weeks after Week 12 [Final Visit])
Population: The Safety (SAF) population included all randomized participants who used at least 1 dose of study drug, including participants who had no post-Baseline assessments unless all dispensed study drug was returned unused.
Measure: Number; unit: Participants
Arm/Group | FMX103 1.5% | Vehicle Foam
Number analyzed (Participants) | 494 | 256
Participants
  All AEs | 98 | 58
  TEAEs | 91 | 54
  Serious TEAEs (SAEs) | 2 | 3
  Participants with any severe TEAE | 1 | 2
  Treatment-related TEAEs | 8 | 7
  AEs leading to study discontinuation | 5 | 2
  TEAEs resulting in death | 0 | 1

ADVERSE EVENTS:
Time Frame: From Day 0/Baseline until the Safety Follow-up (4 weeks after Week 12 [Final Visit])
Arm/Group | FMX103 1.5% | Vehicle Foam
All-Cause Mortality (participants affected / at risk) | 0/494 | 1/256
Serious Adverse Events (participants affected / at risk) | 2/494 | 3/256
Other Adverse Events (participants affected / at risk) | 4/494 | 5/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FMX103 1.5% (N=494) | Vehicle Foam (N=256)
Myocardial infarction (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FMX103 1.5% (N=494) | Vehicle Foam (N=256)
Upper respiratory tract infection (Infections and infestations) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT03142451/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT03142451/SAP_001.pdf